CLINICAL TRIAL: NCT03608085
Title: Community Medication Therapy Management by Pharmacists for Patients Recently Discharged From Heart Failure Hospitalization
Brief Title: Community Pharmacy Medication Therapy Management for Heart Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Providence VA Medical Center (U.S. Federal Agency)
Collaborators: Lifespan (Other); University of Rhode Island (Other)
Responsible Party: Principal Investigator, Tracey H. Taveira, Research Scientist, Providence VA Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1087691-2
Record Dates: First submitted 2018-05-31; First posted 2018-07-31 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Pharmacists

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pharmacist Heart failure MTM training (Experimental): Community pharmacist who will receive heart failure medication therapy management training
  Interventions: Behavioral: Pharmacist Heart failure MTM training
- Patient Heart failure MTM intervention (Experimental): Independently living community dwelling subjects who are prescribed at least 1 cardiovascular medication for HF and 3 additional chronic medications after discharge from the Hospital for an MTM consultation by a pharmacist trained in heart failure medication therapy management.
  Interventions: Behavioral: Patient Heart failure MTM intervention

INTERVENTIONS:
Behavioral: Pharmacist Heart failure MTM training — The MTM training for pharmacists will consist of:
  1. Online material for home self-study (10 contact hours);
  2. Didactic coursework to obtain a national American Pharmaceutical Association (APhA) MTM certification (8 contact hours); and HF pharmacotherapy (4 contact hours);
  3. 1 60-minute sessions of point of care training in the community pharmacy practice lab setting by URI faculty;
  4. Monthly coaching conference calls/webinars with URI and Brown Faculty;
  Other Names: Training intervention for pharmacists
  Arms: Pharmacist Heart failure MTM training
Behavioral: Patient Heart failure MTM intervention — The baseline visit will take place >= 7 but <= 30 days post discharge from the HF hospitalization. Follow-up visits will occur either in person at the patients local pharmacy or via telephone at 30, 60, 90 and 120 days post baseline and will consist of the following:
  Preparation: Develop personal medication record (PMR). Assessment: Medication therapy reconciliation; Education: Review heart failure basics and behavioral goals Planning: Documentation of a medication related action plan and identify medication related problems Implementation: Communication of medication related action plan and changes in heart failure symptoms to the patients providers.
  Follow up: Monitor and evaluate the care plan in collaboration with the patient's providers.
  Other Names: MTM intervention for patients
  Arms: Patient Heart failure MTM intervention

SUMMARY:
Pharmacist-provided medication therapy management (MTM) services have been suggested as a way to improve heart failure (HF) outcomes and counter fragmented care. Nevertheless, broad implementation of MTM services, especially for HF, has not occurred. Therefore, the investigators propose a community engagement pilot study to evaluate the feasibility of 1) training of community pharmacists to perform MTM for HF patients by the University of Rhode Island (URI) Faculty and Brown University Physicians, 2) community pharmacists performing MTM post-training for patients discharged with HF in their own community, 3) establishment of a community based research network (CBRN) and registry to assess the efficacy of the training and the MTM intervention through collaboration among patients with HF, community pharmacists and URI pharmacists and Brown University physicians.

DETAILED DESCRIPTION:
The pharmacists (n=53) of the 20 community pharmacies located in Newport and Bristol Counties will serve as the CBRN intervention sites. The investigators will also enroll 30 independently living community dwelling subjects who are prescribed at least 1 cardiovascular medication for HF and 3 additional chronic medications after discharge from Newport Hospital for an MTM consultation at a CBRN pharmacy. The investigators will assess the implementation of our community intervention based on the REAIM framework. The specific aims are:

Specific Aim 1 (Efficacy): To investigate whether pharmacists who receive the CBRN MTM empowerment training will experience improvement in (aim 1a) self-efficacy and (aim 1b) empowerment from baseline to 180-days.

Specific Aim 2: To assess over the 180-day period, 2a) the reach, 2b) adoption, 2c) implementation (consistency, time spent in lieu of cost and adaptation) including barriers and facilitators.

Specific Aim 3 Exploratory: To determine whether HF patients who receive an MTM intervention from a CBRN community pharmacist experience improvement in HF Self-care behaviors and medication adherence from baseline to 180 days.

Specific Aim 4: To establish a CBRN registry of HF patients to track community pharmacy practices in MTM, hard events such as rehospitalization and death and to evaluate the feasibility of collecting HF outcomes from EPIC electronic health record compared to patient self-report and physician adjudication.

ELIGIBILITY:
Pharmacist Participants:

All pharmacists employed in community pharmacies (n=20) located in either Newport or Bristol county, Rhode Island pharmacies will be offered study enrollment. Pharmacist who meet the inclusion criteria below but chose to not to participate in the training intervention will still be asked to enroll to participate in surveys and interviews to determine their reasons for non-participation.

Inclusion Criteria

* All licensed pharmacists aged ≥18 years that are employed at least part time (minimum of 4 hours per week) in a community pharmacy located in either Newport or Bristol Counties.
* All licensed pharmacists who anticipate working in a community pharmacy located in either Newport or Bristol Counties for the next 6 months
* Able to sign informed consent

The State of Rhode Island pharmacy licensure requirements are as follows:

* Completion of a first professional degree program in pharmacy located within the United States and accredited by the American Council on Pharmaceutical Education.
* Completion of 1,500 internship hours.
* Passage of the North American Pharmacist Licensure Examination (NAPLEX), administered through the National Association of Boards of Pharmacy.
* Passage of the Multistate Pharmacy Jurisprudence Examination (MPJE) for Rhode Island, administered through the National Association of Boards of Pharmacy.

Exclusion Criteria

* Pharmacists with an expired, inactive, suspended license.
* Pharmacist who, in the investigator's opinion, will not comply with study procedures or are unable to provide informed consent.
* Of note, we will not exclude pharmacists who have already completed the general National APhA certification program as this training intervention will focus on MTM in patients with HF

Patient Participants

Thirty patients aged >18 years discharged from Newport Hospital for a HF hospitalization who are prescribed at least 1 cardiovascular medication for HF and at least 3 other medications for chronic disease

Inclusion Criteria

* All subjects >18 years old,
* ≤30 days post-HF hospitalization discharged to a community dwelling,
* Prescribed at least 1 cardiovascular medication for HF (ACE-Inbitors, Angiotensin Receptor Blockers, sacubitril, aldosterone antagonist, diuretics, digoxin, ivabradine and hydralazine, beta blockers and nitrates), and 3 other medications for chronic disease
* Able to sign consent and participate in a MTM consultation

Exclusion Criteria

* Psychiatric instability (acutely suicidal, psychotic) or organic brain injury that precludes self-reporting on health status,
* Discharged to hospice or nursing home or assisted living facilities, or patients with a code status of comfort-measures-only
* Recipients of heart transplant, ventricular assist devices, intravenous inotropic infusions or woman who are pregnant since these conditions would preclude them from standard HF care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Estimated)
Dates: Start 2018-05-23 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in the 31-item MTM self-efficacy scale | baseline to 180 days
  Improvement from baseline in the 31-item MTM Self-efficacy Scale to 180 days. The pharmacists' self-efficacy in performing medication therapy management services scale is a 31-item scale and is divided into the following 5 domains: identify and enroll patients (4 items), provide services (14 items), document and bill services (5 items), collaborating with others (2 items), and specific service tools (8 items). An 11-point Likert scale asks pharmacists to rate "how certain you are that you can do these activities," with response options ranging from 0=cannot do at all to 5=moderately certain can do, and 10= highly certain can do. A total score of ≤124 is determined to represent low self-efficacy, a score of 125-217 is considered moderate, and a score of 218-310 is considered to represent high self-efficacy.

SECONDARY OUTCOMES:
Change in the Conditions of Work Effectiveness Questionnaire II (CWEQ-II Scale) | baseline to 180 days
  Improvement from baseline in (aim 1b) empowerment (Conditions of Work Effectiveness Questionnaire II (CWEQ-II Scale) to 180 days. The Conditions of Work Effectiveness Questionnaire II (CWEQ-II) consists of 19 items that measures the six subscales of structural empowerment (opportunity, information, support, resources, formal power and informal power). These subscales help define the relationship the pharmacist has with the healthcare team and in the practice setting. Based on results of a confirmatory factor analysis that validated the factor structure of this instrument, a total empowerment score is created by summing the six subscales with a score range between 6-30. Responses to all items are made on a 5-point Likert scale (1 = None and 5 = A lot). Total mean scores ranging from 6 to 13 are low levels of empowerment and 14 to 22 are moderate levels of empower and 23 to 30 as high levels of empowerment.

OTHER OUTCOMES:
Reach, adoption and implementation | baseline to 180 days
  The reach, adoption, and implementation will be assessed from baseline to 180-days.
  Reach will be determined by the total number of pharmacists who participate of the total available. Adoption will be determine by the total number of MTM consultations delivered by the community pharmacists from baseline to 180 days.
  To understand facilitators and barriers to the implementation and possibilities of refinement of an MTM training intervention, pre-implementation interviews will be conducted consistent with internal and external environmental domains of the Consolidated Framework of Implementation Research (CFIR) with pharmacists (n=15), HF patients (n=5) and their health care providers (n=5)
Change in heart failure self care behaviors scale (Self Care HF Index v6) | baseline to 180 days
  Change in HF Self-care behaviors (Self Care HF Index v6) scale from baseline to 180 days.
  The HF Self-care Index (v.6) is a 22-item self-administered instrument composed of 3 scales: self-care maintenance, management, and confidence. It addresses diet, exercise, medication use, when to call the health provider, keeping doctor's appointments, weight monitoring, and recognition of change in health status or symptoms. Each scale is scored separately and has a range of 0-100. A score of ≥70 on each scale is considered adequate self-care, though benefit occurs at even lower levels. A score change of half standard deviation (≈8 points) is considered a clinically relevant change.7,8 Our pilot data from the VA hospital showed low self-care scores in HF patients (64.9±19.9) at baseline.
Change in medication adherence | baseline to 180 days
  Adherence to medications will be assessed using pill counts of the cardiovascular medications (ACE-I, ARB, sacubitril, aldosterone antagonist, diuretics, digoxin, ivabradine and hydralazine, beta blockers and nitrates) at baseline and 180-days.
Death and re-hospitalizations | baseline to 180 days
  The total number of and cause of death and re-hospitalizations in patients who receive MTM intervention from a HF MTM trained community pharmacist from baseline to 180 days will be obtained.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Ocean State Research Institute, Providence, Rhode Island
  - Providence VAMC, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: Undecided